CLINICAL TRIAL: NCT03359928
Title: Acute Physiological and Perceptual Responses to Novel Forms of High-intensity Interval Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Naomi Burn, Principal Investigator, Teesside University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 162/17
Record Dates: First submitted 2017-11-16; First posted 2017-12-02 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: High-intensity Interval Exercise; Heart Rate; Rating of Perceived Exertion; Blood Pressure; Acute Mood; Physical Activity Enjoyment
MeSH Terms: interventions — Stair Climbing

STUDY DESIGN:
Intervention Model Description: Using a randomised crossover trial design participants will be randomised computer assisted random sequence generation to sequences in which they are exposed to each experimental condition (exercise modality: stair stepping, stair climbing and non-contact boxing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Boxing (Experimental): In each of the three sessions a different exercise modality will be conducted, in a randomised sequence. Non-contact boxing involves boxing "punch pads" that will be held by the one of the researchers, while wearing protective boxing gloves. Each exercise modality will be conducted following a high-intensity interval protocol (4 x 60 seconds of exercise interspersed with 60 seconds of rest). During each exercise bout participants will be encouraged to exercise at an intensity that elicits a heart rate of ≥85% of maximum, which will always be followed by 60 seconds of passive recovery. Participants will complete a 5 minute warm-up and a 2 minute cool down and stretch after the exercise bouts have been completed.
  Interventions: Behavioral: Boxing
- Stair stepping (Experimental): Participants will complete 3 sessions of exercise. In each of the three sessions a different exercise modality will be conducted in a randomised sequence. Stair stepping involves stepping on to and off a 35 cm Reebok exercise bench, repeatedly. Each exercise modality will be conducted following a high-intensity interval protocol (4 x 60 seconds of exercise interspersed with 60 seconds of rest). During each exercise bout participants will be encouraged to exercise at an intensity that elicits a heart rate of ≥85% of maximum, which will always be followed by 60 seconds of passive recovery. Participants will complete a 5 minute warm-up and a 2 minute cool down and stretch after the exercise bouts have been completed.
  Interventions: Behavioral: Stair stepping
- Stair climbing (Experimental): In each of the three sessions a different exercise modality will be conducted, in a randomised sequence. Stair climbing involves continuously ascending the stairs located in a public access staircase. Each exercise modality will be conducted following a high-intensity interval protocol (4 x 60 seconds of exercise interspersed with 60 seconds of rest).
  During each exercise bout participants will be encouraged to exercise at an intensity that elicits a heart rate of ≥85% of maximum, which will always be followed by 60 seconds of passive recovery. Participants will complete a 5 minute warm-up and a 2 minute cool down and stretch after the exercise bouts have been completed.
  Interventions: Behavioral: Stair climbing

INTERVENTIONS:
Behavioral: Boxing — as already discussed
  Arms: Boxing
Behavioral: Stair stepping — as already discussed
  Arms: Stair stepping
Behavioral: Stair climbing — as already discussed
  Arms: Stair climbing

SUMMARY:
Randomised cross-over study seeking to explore the acute physiological and perceptual responses to three novel forms of high-intensity interval training (HIT).

DETAILED DESCRIPTION:
Randomised cross-over study seeking to explore the acute physiological (heart rate and blood pressure) and perceptual responses (rating of perceived exertion, mood and enjoyment) to three novel forms (non-contact boxing, stair stepping and stair climbing) of high-intensity interval training (HIT).

ELIGIBILITY:
Inclusion Criteria:

* adult (≥18 years) employees
* no health conditions that preclude them from exercise and on no medication, information obtained via their self-report.
* able to understand written and spoken English.
* participants reporting that they are asthmatic will allowed to participate with medical clearance and instructed to bring their bronchodilator medication and use it when required.

Exclusion Criteria:

* symptoms of or known presence of heart disease
* condition or injury or co-morbidity affecting the ability to undertake exercise
* diabetes mellitus
* early family history of sudden cardiac death
* pregnancy or likelihood of pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Heart rate | 6 months
  Second-to-second heart rate monitoring throughout exercise sessions using wrist worn Polar A360 heart rate monitors

SECONDARY OUTCOMES:
Mood | 6 months
  Acute mood state
Enjoyment | 6 months
  Physical activity enjoyment scale (PACES). Range of possible scores from 18-126, higher scores indicate higher enjoyment.
RPE | 6 months
  Rating of perceived exertion
Blood pressure | 6 months
  Measured using automatic blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weston, PhD, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No